CLINICAL TRIAL: NCT03322540
Title: A Phase 2, Randomized, Double-Blind Study of Pembrolizumab (MK-3475) Plus Epacadostat (INCB024360) Versus Pembrolizumab Plus Placebo as First-Line Treatment in Patients With Metastatic Non-Small Cell Lung Cancer Expressing High Levels of PD-L1
Brief Title: Pembrolizumab Plus Epacadostat vs Pembrolizumab Plus Placebo in Metastatic Non-Small Cell Lung Cancer (KEYNOTE-654-05/ECHO-305-05)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KEYNOTE-654-05/ECHO-305-05; 2017-001841-28 (EudraCT Number)
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; programmed cell death 1 (PD-1) inhibitor; indoleamine 2; 3-dioxygenase 1 (IDO1) inhibitor
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; epacadostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: With the implementation of Amendment 05 the study is no longer blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Epacadostat (Experimental): Participants received pembrolizumab 200 mg as an intravenous (IV) infusion, every three weeks (Q3W) starting on Day 1 of each cycle for up to 35 administrations in combination with epacadostat 100 mg orally, twice daily. Epacodostat administration was discontinued after the implementation of protocol amendment 05.
  Interventions: Drug: Pembrolizumab; Drug: Epacadostat
- Pembrolizumab + Placebo (Active Comparator): Participants received pembrolizumab 200 mg by IV infusion, Q3W starting on Day 1 of each cycle for up to 35 administrations in combination with matching placebo orally, twice daily. Placebo administration was discontinued after the implementation of protocol amendment 05.
  Interventions: Drug: Pembrolizumab; Drug: Placebo

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab administered intravenously every 3 weeks.
  Other Names: MK-3475
Drug: Epacadostat — Epacadostat administered orally twice daily.
  Other Names: INCB024360
  Arms: Pembrolizumab + Epacadostat
Drug: Placebo — Matching placebo administered orally twice daily.
  Arms: Pembrolizumab + Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pembrolizumab plus epacadostat compared to pembrolizumab plus placebo as first-line treatment in participants with metastatic non-small cell lung cancer (NSCLC) expressing high levels of programmed cell death ligand 1 (PD-L1).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of stage IV NSCLC without epidermal growth factor receptor (EGFR)-sensitizing mutation, ROS1 and/or anaplastic lymphoma kinase (ALK) translocation.
* Measurable disease based on RECIST 1.1.
* Tumor tissue that demonstrates programmed cell death ligand 1 (PD-L1) expression in ≥ 50% of tumor cells (tumor proportion score [TPS] ≥ 50%) as assessed by immunohistochemistry at a central laboratory.
* Life expectancy of at least 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function per protocol-defined criteria.

Exclusion Criteria:

* Known untreated central nervous system metastases and/or carcinomatous meningitis.
* History of (noninfectious) pneumonitis that required systemic steroids or current pneumonitis/interstitial lung disease.
* Symptomatic ascites or pleural effusion.
* Known history of an additional malignancy, except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy.
* Active autoimmune disease that has required systemic treatment in past 2 years.
* Has had an allogeneic tissue/solid organ transplant.
* Has a known history of human immunodeficiency virus (HIV) infection. HIV testing is not required unless mandated by the local health authority.
* Has known history of or is positive for active Hepatitis B (HBsAg reactive) or has active Hepatitis C (HCV RNA). Note: Testing must be performed to determine eligibility.
* History or presence of an abnormal electrocardiogram (ECG) that, in the Investigator's opinion, is clinically meaningful.
* Use of protocol-defined prior/concomitant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2020-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, MD, Study Director — Incyte Corporation
Locations (101):
- United States (15):
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Innovative Clinical Research Institute, Whittier, California
  - Florida Cancer Specialists (South Region), Fort Myers, Florida
  - Florida Cancer Specialists (North Region), St. Petersburg, Florida
  - Southeastern Regional Medical Center, Inc., Newnan, Georgia
  - Anne Arundel Health System Research Institute, Annapolis, Maryland
  - Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - Maryland Oncology Hematology, P.A., Rockville, Maryland
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Minnesota Oncology Hematology, PA, Coon Rapids, Minnesota
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Tennessee Oncology, PLLC/The Sarah Cannon Research Institute, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC/The Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology-South Austin, Austin, Texas
- Australia (2):
  - Austin Health-Austin Hospital, Heidelberg, Victoria
  - St John of God Murdoch Medical Clinic, Murdoch, Western Australia
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - Moncton Hospital - Horizon Health Network, Moncton, New Brunswick
  - William Osler Health System, Brampton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Sault Area Hospital, Sault Ste. Marie, Ontario
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - Regionshospitalet Herning, Herning
  - Odense Universitetshospital, Odense
- SA Tartu Ulikooli Kliinikum, Tartu, Estonia
- Ireland (2):
  - Galway University Hospital, Galway, Connacht
  - St Vincents University Hospital, Dublin
- Israel (5):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (2):
  - IRCCS A.O.U. San Martino - IST, Genova
  - Policlinico Universitario Agostino Gemelli, Roma
- Japan (17):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kurume University Hospital, Kurume, Fukuoka
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - Shizuoka Cancer Center, Nagaizumi-chō, Shizuoka
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - National Cancer Center Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Wakayama Medical University Hospital, Wakayama
- Malaysia (5):
  - Institut Kanser Negara - National Cancer Institute, Putrajaya, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - University Malaya Medical Centre, Kuala Lumpur
  - Pantai Hospital Kuala Lumpur, Kuala Lumpur
  - Sarawak General Hospital, Kuching
- Poland (8):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka, Bydgoszcz
  - Centrum Onkologii. Instytut im. Marii Sklodowskiej-Curie, Gliwice
  - Swietokrzyskie Centrum Onkologii SPZOZ, Kielce
  - Przychodnia Lekarska Komed, Konin
  - Samodzielny Publiczny Zespol Gruzlicy i Chorob Pluc, Olsztyn
  - Wojewodzki Szpital im. Zofii z Zamoyskich Tarnowskiej w Tarnobrzegu, Tarnobrzeg
  - Centrum Onkologii-Instytut im. Marii Sklodowskiej-Curie, Warsaw
  - Swietokrzyskie Centrum Onkologii SPZOZ, Kielce, Świętokrzyskie Voivodeship
- Russia (6):
  - Belgorod Regional Oncology Dispensary, Belgorod
  - Central Clinical Hospital with polyclinic, Moscow
  - Moscow Research Oncology Institute named after P.A. Hertsen, Moscow
  - SBHI Leningrad Regional Clinical Hospital, Saint Petersburg
  - SBHI Samara Regional Clinical Oncology Dispensary, Samara
  - Republican Clinical Oncology Dispensary of Republic of Bashkortostan, Ufa
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Gacheon University Gil Medical Center, Incheon
- Spain (7):
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital General de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico de Valencia, Valencia
- Switzerland (5):
  - Oncological Institute of Southern Switzerland, Bellinzona
  - Inselspital Universitatsspital Bern, Bern
  - Hopitaux Universitaires de Geneve HUG., Geneva
  - Kantonsspital Winterthur, Winterthur
  - Universitaetsspital Zuerich, Zurich
- Turkey (Türkiye) (5):
  - Basken Uni. Adana Dr.Turgut Noyan Uygulama ve Arastirma Merkezi, Adana
  - Ankara University Medical Faculty, Ankara
  - Akdeniz Universitesi Tip Fakultesi, Antalya
  - Erciyes Universitesi Tip Fakultesi, Kayseri
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi Hastanesi, Konya
- Ukraine (9):
  - MI Kryviy Rih Center of Dnipropetrovsk Regional Council, Kryvyi Rih, Dnipropetrovsk Oblast
  - Dnipropetrovsk City Multidiscipline Clinical Hosp.4 of DRC, Dnipropetrovsk
  - Grigoriev Institute for medical Radiology NAMS of Ukraine, Kharkiv
  - PP PPC Acinus Medical and Diagnostic Centre, Kirovohrad
  - Kyiv City Clinical Oncological Center, Kyiv
  - Dobryi Prognoz, Kyiv
  - Volyn Regional Oncological Dispensary, Lutsk
  - MI Odessa Regional Oncological Centre, Odesa
  - Zaporizhzhya Regional Clinical Oncology Center, Zaporizhzhya
- Leeds Teaching Hospital NHS Trust. St. James University Hospital, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tokito T, Kolesnik O, Sorensen J, Artac M, Quintela ML, Lee JS, Hussein M, Pless M, Paz-Ares L, Leopold L, Daniel J, Munteanu M, Samkari A, Xu L, Butts C. Epacadostat plus pembrolizumab versus placebo plus pembrolizumab as first-line treatment for metastatic non-small cell lung cancer with high levels of programmed death-ligand 1: a randomized, double-blind phase 2 study. BMC Cancer. 2024 Jul 25;23(Suppl 1):1251. doi: 10.1186/s12885-023-11203-8. PMID 39054476

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 154 participants were randomized in 1:1 to either combination (Pembrolizumab+Epacadostat) and control (Pembrolizumab+Placebo) groups. As of Amendment 05, study design was changed to unblinded, open-label, and single-arm (epacadostat and placebo were removed).
Pre-assignment Details: Phase 3 design of the study has been amended soon after it had started to a prospectively randomized phase 2 study. At the time of amendment existing participants were given a choice to move/participate in the new phase 2 study, and some participants who chose to discontinue the study at phase 3 were assigned to "study terminated by sponsor" as the reason for not completing the study in disposition table. The results posted are combined in the prospectively redesigned phase 2 trial.
Period: Overall Study
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab + Placebo
Started | 77 | 77
Number of Subjects Received Treatment (Actual Treatment) (ASaT) | 75 | 77
Completed | 46 | 40
Not Completed | 31 | 37
Not completed — Death | 21 | 28
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 7 | 6
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Study terminated by sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab + Placebo | Total
Number analyzed (Participants) | 77 | 77 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (9.5) | 66.9 (10.1) | 65.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 42
  Male | 53 | 59 | 112
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 25 | 23 | 48
  White | 52 | 54 | 106
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic Or Latino: Hispanic Or Latino | 7 | 4 | 11
  Not Hispanic Or Latino: Not Hispanic Or Latino | 66 | 73 | 139
  Not Hispanic Or Latino: Not Reported | 3 | 0 | 3
  Not Hispanic Or Latino: Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) of Pembrolizumab Plus Epacadostat Versus Pembrolizumab Plus Placebo
Description: ORR is defined as the proportion of participants who have a confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 based on blinded independent central review (BICR).
Time Frame: Up to approximately 6 months
Population: ITT population consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab + Placebo
Number analyzed (Participants) | 77 | 77
percentage of participants | 32.5 [22.2 to 44.1] | 39.0 [28.0 to 50.8]
Statistical Analysis 1: Comparison: Pembrolizumab + Epacadostat vs Pembrolizumab + Placebo; Test type: Superiority; p = 0.8000, Stratified Miettinen and Nurminen method; One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in Percentages = -6.5, 95% CI 2-sided [-21.5 to 8.7] — Point estimate was assessed based on Miettinen & Nurminen method stratified by predominant tumor histology (squamous vs non-squamous)

2. Secondary Outcome: Progression-free Survival (PFS) of Pembrolizumab + Epacadostat Versus Pembrolizumab + Placebo
Description: PFS is defined as the time from randomization to the first documented progressive disease per RECIST v1.1 based on BICR or death due to any cause, whichever occurs first.
Time Frame: Up to approximately 36 months
Population: ITT population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab + Placebo
Number analyzed (Participants) | 77 | 77
months | 6.7 [4.3 to 8.2] | 6.2 [4.3 to NA] — Upper bound was not estimable

3. Secondary Outcome: Overall Survival (OS) of Pembrolizumab + Epacadostat Versus Pembrolizumab + Placebo
Description: OS is defined as the time from randomization to death due to any cause.
Time Frame: Up to approximately 36 months
Population: ITT population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pembrolizumab + Epacodostat: Participants received pembrolizumab 200 mg as an intravenous (IV) infusion, every three weeks (Q3W) starting on Day 1 of each cycle for up to 35 administrations in combination with epacadostat 100 mg orally, twice daily. Epacodostat administration was discontinued after the implementation of protocol amendment 05.
Arm/Group | Pembrolizumab + Epacodostat | Pembrolizumab + Placebo
Number analyzed (Participants) | 77 | 77
Months | NA [NA to NA] — Median Overall Survival was not reached | NA [NA to NA] — Median Overall Survival was not reached

4. Secondary Outcome: Duration of Response (DOR) of Pembrolizumab + Epacadostat Versus Pembrolizumab + Placebo
Description: DOR is defined as the time from the earliest date of qualifying response until earliest date of disease progression per RECIST v1.1 or death from any cause, whichever comes first.
Time Frame: Up to approximately 36 months
Population: DOR included all responders in ITT population. Response duration was calculated from product-limit (Kaplan-Meier) method for censored data.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab + Epacodostat | Pembrolizumab + Placebo
Number analyzed (Participants) | 77 | 77
Months | 6.2 [1.9 to 6.5] | NA [1.9 to 8.6] — Median was not reached in this arm.

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: AE is defined as any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: Up to 37 months
Measure: Number; unit: Participants
Arm/Group | Pembrolizumab + Epacodostat | Pembrolizumab + Placebo
Number analyzed (Participants) | 75 | 77
Participants | 72 | 72

6. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to AEs
Description: as for outcome 5
Time Frame: Up to 37 months
Measure: Number; unit: Participants
Arm/Group | Pembrolizumab + Epacodostat | Pembrolizumab + Placebo
Number analyzed (Participants) | 75 | 77
Participants | 15 | 12

ADVERSE EVENTS:
Time Frame: Up to 37 months
Description: The all participants as treated (APaT) population will be used for the analysis of safety data in this study. The APaT population consists of all randomized participants who received at least one dose of study treatment.
Groups:
- Total: Total
Arm/Group | Pembrolizumab + Epacadostat | Pembrolizumab + Placebo | Total
All-Cause Mortality (participants affected / at risk) | 23/75 | 29/77 | 52/152
Serious Adverse Events (participants affected / at risk) | 36/75 | 35/77 | 71/152
Other Adverse Events (participants affected / at risk) | 69/75 | 67/77 | 136/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Epacadostat (N=75) | Pembrolizumab + Placebo (N=77) | Total (N=152)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Autoimmune myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Cholangitis sclerosing (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Fear of death (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
High-grade B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 2 (2)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 8 (8) | 14 (14)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 2 (3)
Pneumonia (Infections and infestations) | 6 (6) | 7 (7) | 13 (13)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 6 (6)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Priapism (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Pseudodiverticular disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Tumour pseudoprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Epacadostat (N=75) | Pembrolizumab + Placebo (N=77) | Total (N=152)
Alanine aminotransferase increased (Investigations) | 5 (5) | 5 (8) | 10 (13)
Amylase increased (Investigations) | 8 (9) | 4 (8) | 12 (17)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 10 (12) | 17 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (22) | 10 (12) | 27 (34)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 4 (7) | 8 (11)
Asthenia (General disorders) | 8 (9) | 6 (8) | 14 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (13) | 8 (11) | 18 (24)
Blood creatinine increased (Investigations) | 4 (4) | 7 (8) | 11 (12)
Chest pain (General disorders) | 5 (5) | 6 (7) | 11 (12)
Chills (General disorders) | 4 (5) | 1 (2) | 5 (7)
Constipation (Gastrointestinal disorders) | 20 (23) | 18 (21) | 38 (44)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 8 (8) | 15 (17)
Decreased appetite (Metabolism and nutrition disorders) | 17 (18) | 10 (12) | 27 (30)
Diarrhoea (Gastrointestinal disorders) | 16 (30) | 17 (25) | 33 (55)
Dizziness (Nervous system disorders) | 5 (5) | 6 (6) | 11 (11)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4) | 9 (9)
Dysgeusia (Nervous system disorders) | 4 (4) | 1 (1) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 10 (13) | 20 (26)
Fatigue (General disorders) | 9 (11) | 16 (21) | 25 (32)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7) | 13 (13)
Headache (Nervous system disorders) | 13 (15) | 4 (4) | 17 (19)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (7) | 2 (2) | 8 (9)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (5) | 7 (11) | 9 (16)
Hyperthyroidism (Endocrine disorders) | 8 (8) | 6 (6) | 14 (14)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6) | 5 (7) | 9 (13)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (8) | 1 (1) | 7 (9)
Hypotension (Vascular disorders) | 2 (2) | 4 (4) | 6 (6)
Hypothyroidism (Endocrine disorders) | 10 (11) | 6 (6) | 16 (17)
Insomnia (Psychiatric disorders) | 6 (7) | 4 (5) | 10 (12)
Lipase increased (Investigations) | 9 (9) | 4 (5) | 13 (14)
Lymphocyte count decreased (Investigations) | 1 (1) | 4 (7) | 5 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (9) | 9 (11)
Nasopharyngitis (Infections and infestations) | 2 (2) | 8 (10) | 10 (12)
Nausea (Gastrointestinal disorders) | 14 (16) | 8 (8) | 22 (24)
Oedema peripheral (General disorders) | 4 (6) | 5 (5) | 9 (11)
Oral candidiasis (Infections and infestations) | 2 (3) | 4 (6) | 6 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (4) | 9 (10)
Pneumonia (Infections and infestations) | 4 (4) | 3 (3) | 7 (7)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 16 (21) | 16 (22) | 32 (43)
Pyrexia (General disorders) | 7 (8) | 8 (8) | 15 (16)
Rash (Skin and subcutaneous tissue disorders) | 15 (22) | 11 (16) | 26 (38)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5) | 7 (8) | 11 (13)
Respiratory tract infection (Infections and infestations) | 5 (5) | 1 (2) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 8 (8) | 14 (14)
Urinary tract infection (Infections and infestations) | 4 (4) | 6 (10) | 10 (14)
Vomiting (Gastrointestinal disorders) | 7 (8) | 6 (6) | 13 (14)
Weight decreased (Investigations) | 7 (7) | 8 (8) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT03322540/Prot_001.pdf
  • Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT03322540/SAP_002.pdf